CLINICAL TRIAL: NCT01479192
Title: Breast Cancer Prevention With Fenretinide in Young Women at Genetic and Familil Risk. A Phase III Randomized Clinical Trial
Brief Title: Fenretinide in Healthy Young Women at Genetic and Familial Risk
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: very low rate of patient accrual
Sponsor: European Institute of Oncology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: IEO S462/109; 2009-010260-41 (EudraCT Number)
Record Dates: First submitted 2011-11-22; First posted 2011-11-24 (Estimated); Last update posted 2018-11-07 (Actual); Status verified 2015-12

CONDITIONS: High-Risk Cancer
Keywords: breast; cancer; prevention; fenretinide
MeSH Terms: conditions — Neoplasms | interventions — Fenretinide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Fenretinide (Experimental): 100mg: 2cps/day for 5 years followed by
  Interventions: Drug: Fenretinide
- Placebo (Placebo Comparator): matched placebo 2 cps/day for 5 years
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Fenretinide — 100mg (2cps/day) for 5 years
  Arms: Fenretinide
Other: Placebo — 2 cpr/day of matched placebo for 5 years
  Arms: Placebo

SUMMARY:
The purpose of this trial is to assess the effect of fenretinide (4-HPR), a vitamin A derivative, in reducing the incidence of breast cancer in healthy premenopausal women at increased familial/genetic risk for breast cancer

DETAILED DESCRIPTION:
Retinoids have been studied as chemo preventive compounds in clinical trials because of their acknowledged role in regulating cell growth, differentiation and apoptosis in preclinical models. Induction of apoptosis is a unique feature of fenretinide (4-hydroxyphenylretinamide, 4-HPR),(2) the most widely studied retinoid in clinical trials of breast cancer chemoprevention for its selective accumulation in the breast tissue and its very low toxicity. The fifteen-year follow up of a randomized phase III trial of fenretinide to prevent second breast cancer indicates that fenretinide induced a 17%, durable reduction of second breast cancer incidence. When stratified by menopausal status, the analysis showed a 38%, statistically significant reduction of second breast cancers in premenopausal women and this protective effect persisted for up to 15 years, i.e. 10 years after treatment cessation. Importantly, the younger were the women, the greater was the trend of benefit of fenretinide, with a remarkable 50% risk reduction in women aged 40 years or younger, whereas the benefit disappeared after age 55. One explanation for the different effects of fenretinide according to menopausal status or age is a different modulation of circulating IGF-I in premenopausal and postmenopausal women, with a reduction of IGF-I levels only in premenopausal subjects.

When considering the protective activity of fenretinide on second breast cancer in young women and a similar trend on ovarian cancer (the latter at least during intervention)(4, 5), it appears that young women at high risk such as those with germ line BRCA-1 and 2 mutations or those with a high family risk may be ideal candidates for further investigation on this retinoid. Indeed, fenretinide is highly effective in inhibiting the growth of BRCA-1 mutated breast cancer cell lines. Since a reduction of second breast cancer might be a surrogate marker of primary prevention, a favourable effect of fenretinide provides strong rationale for a primary prevention trial in unaffected women at high-risk for breast cancer.

Importantly, at clinically relevant doses, fenretinide has shown to induce NO-mediated apoptosis in human and murine BRCA-1 mutated cancer cells, and In this ability fenretinide was the most potent of the phenylretinamide analogues against BRCA-1 mutated breast cancer cells.

Additionally, recent studies have shown that 4-HPR modulates gene expression in ovarian cells, with an up-regulation of expression of proapoptotic genes in OVCA433 cells and down-regulation of mutant BRCA genes in IOSE (premalignant) cells and OVCA433 cells. This suggests a preventive effect in premalignant cells and a treatment effect in cancer cells.

Increasing evidence sustains a link between the rising prevalence of metabolic syndrome in the Western world and breast cancer incidence. The retinol-binding protein 4 (RBP4), an adipocyte-secreted molecule, is the only specific transport protein for retinol in the blood and correlates with components of the metabolic syndrome, including increased body-mass index, waist-to-hip ratio, serum triglycerides. Plasma concentrations of RBP4 are known to decrease proportionally with retinol during fenretinide administration and normalization of RBP4 by fenretinide in insulin-resistant obese mice has shown to improve insulin action and glucose tolerance.

Among other molecular biomarker candidates for malignant tumours, cell-free DNA circulating in serum is very promising. Unlike uniformly truncated DNA released from apoptotic cells, DNA released from dead cancer cells varies in size. Serum DNA integrity and the ratio of longer fragments to total DNA may be clinically useful for detecting breast cancer progression. Since free-circulating DNA is a non-invasive approach and can be detected in cancer patients and not in disease-free individuals, it will be interesting to study if it can be used as an early detection biomarker.

Breast cancer chemoprevention is rapidly evolving, and there is strong evidence that primary chemoprevention is possible. The more established preventive agents so far are SERMs (selective estrogen receptor modulators), while AIs (aromatase inhibitors) are currently under investigation in postmenopausal populations. All these drugs involve directly the hormonal pathway of the pathogenesis of the disease, and their target is most likely limited to hormone responsive tumours. Tamoxifen has great effect as a chemo preventive agent but it may have serious side effects, while raloxifene may have a better toxicity profile, especially as concerns the risk of endometrial cancer, but it has been tested only in post menopause. Fenretinide has shown to possess several good properties both in preclinical models and clinical trials. In particular, the prolonged effect demonstrated in the phase III trial chemopreventive trial in breast cancer subjects, together with a trend of protective effect on the ovaries, has been accompanied by a very low toxicity profile (mainly reversible skin dryness and rashes and dark adaptation difficulties, often overcome by a monthly weekend suspension of the drug).

All these characteristics make fenretinide an excellent candidate for chemoprevention in a cohort of young healthy women with a high susceptibility to early onset breast and ovarian cancer, such as those who carry a BRCA 1/2 mutation or have a significant family risk. Since the drug activities are probably not strictly influenced by hormonal responsiveness, it is possible that it may have effect also on hormone non-responsive cancers, and this may be very useful particularly in case of BRCA1 mutation carriers.

Side effects and toxicity: visual symptoms (diminished dark adaptability, dryness and lacrimation) have been reported in approximately 20% of subjects. These symptoms may occur more frequently at the start of intervention and they tend to recover with time often without the need for treatment discontinuation. A regular three-days/month drug suspension has been adopted for a long time in clinical studies to minimize visual impairment. Although this side effect is in many women manageable (especially following the regular three day suspension) and reversible, it must be remembered that the dark adaptability impairment might be potentially dangerous in certain situations such as driving from the bright sun into a dark tunnel or night driving.

Dermatological disorders, such as skin and mucosal dryness, pruritus and urticaria can be detected in about 18% of subjects. Mild gastrointestinal symptoms are reported in around 13% of patients. Interestingly, with the exception of ocular surface disorders, the incidence of the other adverse effects seems to decrease with time and is significantly more frequent in postmenopausal women.

Liver toxicity and increase in blood lipid levels, especially triglycerides, are reported but not consistently in the literature.

Like other retinoids, fenretinide may be potentially teratogenic, although available studies show no genotoxic effects in vitro and in vivo, and a lack of storage in the human embryo.

Thus, appropriate measures of contraception should be adopted when treating potentially fertile women.

ELIGIBILITY:
Inclusion Criteria:

1. 20-46 years old women with a known BRCA ½ mutation or with a risk of being a mutation carrier ≥20%.
2. Performance status =0
3. Willingness to avoid pregnancy during treatment and 12 months after drug cessation
4. No clinical and radiological evidence of breast cancer and ovarian disease
5. Signed informed consent

Exclusion Criteria:

1. History of breast cancer or any other malignancy with the exclusion of CIN and non-melanoma skin cancer
2. Child bearing or breast feeding
3. Genetic test result (BRCA)=true negative
4. Blood test alterations (grade ≥2 based on the NCI Common Toxicity Criteria)
5. Previous or concurrent use of SERMs, e.g. tamoxifen (for more than 12 months; if less, a two-months wash-out is required before entering the study)
6. Severe psychiatric disorders or inability to comply to the protocol procedures
7. Any other factor that, at the investigator's discretion, contraindicates the use of fenretinide

Ages: 20 Years to 46 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2009-12; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Breast cancer incidence | every 6 months for 15 years
  The aim of the proposed trial is to assess the efficacy of fenretinide, (4 hydroxyphenilretinamide, 4-HPR), a vitamin A derivative, in reducing the incidence of breast cancer (BC) in healthy young premenopausal women at increased familial/genetic risk for BC (i.e. BRCA1 or BRCA2 mutation carriers or subjects at high risk of being carriers). The primary endpoint is the incidence of invasive BC and ductal intraepithelial neoplasia (DIN), histologically diagnosed.

SECONDARY OUTCOMES:
Incidence of other non-invasive breast disorders, ovarian cancers and other cancers. | every 6 months for 15 years
  Incidence of other non-invasive breast disorders, ovarian cancers and other cancers.
  Early intermediate biomarkers of efficacy after 12, 36, and 60 months of treatment. We will also evaluate the percent change in circulating biomarkers of the IGF system, androgens, retinol binding protein (RBP-4), insulin, blood glucose and VEGF, after 12, 36 and 60 months of treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Umberto Veronesi, Study Chair — European Institute of Oncology
Locations (1):
- European Institute of Oncology, Milan, Italy